CLINICAL TRIAL: NCT05584761
Title: A Perspective, Multicenter, Open-label and Observational Trial for Unrelated Umbilical Cord Blood Stem Cell Microtransplantation Combined With Azacitidine Based Treatment for Advanced MDS,CMML-2 and Secondary AML.
Brief Title: Unrelated Umbilical Cord Blood Stem Cell Combined With Azacitidine Based Treatment for Advanced MDS,CMML-2 and sAML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-271
Record Dates: First submitted 2022-10-06; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia-2; Secondary Acute Myeloid Leukemia
Keywords: umbilical cord blood stem cell; microtransplantation; myelodysplastic syndromes; Chronic myelomonocytic leukemia; secondary acute myeloid leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): unrelated umbilical cord blood stem cell microtransplantation combined with AZA/AZA+ based treatment.
  A single unit of unrelated umbilical cord blood was reinfused within 24-72 hours after the end of AZA or chemotherapy, and the longest delay was 96 hours after the end of chemotherapy. The umbilical cord blood was matched at 0-3/10 locus.
  Specific treatment options:
  1. AZA monotherapy:
     Azacitidine 75mg·m-2·d-1, d1-d7, subcutaneous injection;
  2. VA :
     Azacitidine 75mg·m-2·d-1, d1-d7, subcutaneous injection; Venetoclax (VEN) 100mg d1,200mg d2,400mg d3 to d14, orally.
  3. VAH:
  Azacitidine 75mg·m-2·d-1, d1-d7, subcutaneous injection; Venetoclax (VEN) 100mg d1, 200mg d2,400mg d3 to d14, orally. Homoharringtonine injection (HHT) 2-3mg d1 to d14 was intravenously injected. During the period, the medication time was adjusted according to the patient's blood condition and complications
  Interventions: Drug: unrelated umbilical cord blood

INTERVENTIONS:
Drug: unrelated umbilical cord blood — A single unit of unrelated umbilical cord blood was reinfused within 24-72 hours after the end of AZA or chemotherapy, and the longest delay was 96 hours after the end of chemotherapy. The umbilical cord blood was matched at 0-3/10 locus.
  Microtransplantation of umbilical cord blood: single unit of unrelated cord blood (HLA 0-5/10 or 0-3/6 matched, TNC 1-2×107/Kg body weight), AZA or homoharringtonine infusion 24-72 hours after the end of injection.

SUMMARY:
This research is being done to study the efficacy and safety of unrelated umbilical cord blood stem cell microtransplantation combined with azacitidine(AZA) based treatment for advanced myelodysplastic syndromes(MDS), Chronic myelomonocytic leukemia-2(CMML-2) and secondary acute myeloid leukemia(sAML). The study protocol involved unrelated umbilical cord blood stem cell combined with azacitidine based treatment, which including azacitidine alone and azacitidine plus a targeted agent or chemotherapy agent.

DETAILED DESCRIPTION:
This is a perspective, multicenter, open-label and observational trial for unrelated umbilical cord blood stem cell microtransplantation combined with azacitidine based treatment for advanced MDS,CMML-2 and secondary AML. The study protocol is AZA /AZA+ combined with umbilical cord blood stem cell microtransplantation for patients who met the inclusion criteria in higher-risk MDS(HR-MDS), CMML and sAML.

Demethylating agents are mainly decitabine (DAC) and azacitidine (AZA), both of which have been approved by the FDA for the treatment of MDS. The FDA has also approved hypomethylating agents for the treatment of CMML.Secondary acute myeloid leukemia (sAML) refers to acute myeloid leukemia with progression from a preexisting hematologic disease, such as myelodysplastic syndrome (MDS) or myeloproliferative disorder (MPN) (excluding chronic myelomonocytic leukemia). Currently, there is no standard treatment for sAML. Based on the results of retrospective studies and clinical trials, the efficacy of hypomethylating agents in the treatment of sAML is not weaker than that of traditional intensive induction therapy and other reduced-intensity therapy or best supportive care.

The development of microtransplantation has provided new treatment modalities in patients who are not candidates for conventional allogeneic hematopoietic stem cell transplantation. In China, Huisheng Ai team proposed the concept of micro-transplantation. Micro-transplantation (MST) is a new concept and method that combines conventional chemotherapy or targeted drugs with allogeneic stem cell infusion. Microtransplantation is combined with infusion of G-CSF mobilized peripheral blood stem cells (G-PBSC) from HLA-mismatched donors on the basis of killing leukemia cells by chemotherapy or targeted drugs. Thus, donor microchimerism (donor cells <1-5%) can be formed to induce donor/recipient anti-leukemia (GVL/RVL) effect and promote hematopoietic recovery in recipients without full donor engraftment and almost no risk of GVHD. The clinical results have also been verified in several research centers in the United States, Australia, Spain and other countries, which show that micro-transplantation technology can promote hematopoietic recovery, produce graft-versus-tumor effect and recipientversus-tumor effect, and provide a new safe and effective treatment method for the treatment of hematological diseases and solid tumors.

Participants will receive unrelated umbilical cord blood transfusion during at least 1-2 cycles of treatment.The specific process is as follows:

A single unit of unrelated umbilical cord blood was reinfused within 24-72 hours after the end of AZA or chemotherapy, and the longest delay was 96 hours after the end of chemotherapy. The umbilical cord blood was matched at 0-3/10 locus.

Specific treatment options:

1. AZA monotherapy:

   Azacitidine 75mg·m-2·d-1, d1-d7, subcutaneous injection;
2. VA :

   Azacitidine 75mg·m-2·d-1, d1-d7, subcutaneous injection; Venetoclax (VEN) 100mg d1,200mg d2,400mg d3 to d14, orally.
3. VAH :

Azacitidine 75mg·m-2·d-1, d1-d7, subcutaneous injection; Venetoclax (VEN) 100mg d1, 200mg d2,400mg d3 to d14, orally. Homoharringtonine injection (HHT) 2-3mg d1 to d14 was intravenously injected. During the period, the medication time was adjusted according to the patient's blood condition and complications If severe adverse reactions (such as grade 3 or above infection and bone marrow suppression) occurred, the next course of treatment was postponed according to the situation.

Microtransplantation of umbilical cord blood: single unit of unrelated cord blood (HLA 0-5/10 or 0-3/6 matched, TNC 1-2×107/Kg body weight), AZA or homoharringtonine infusion 24-72 hours after the end of injection.

It is expected that about 50 patients will take part in this research study.

ELIGIBILITY:
1. MDS patients diagnosed due to bone marrow morphology and immunophenotyping (met the World Health Organization(WHO) 2016 diagnosis criterion) and met revised the International Prognostic Scoring System(IPSS) prognostic risk categories intermediate(>3-≤4.5), high(>4.5-≤6), and very high risk(>6), or CMML-2(PB 5-19% or bone marrow 10-19% blast equivalent, and/or when any Auer rods are present) patients diagnosed due to bone marrow morphology and immunophenotyping (met the WHO 2016 diagnosis criterion) with white blood cell count(WBC)<13x109/L, or AML patients diagnosed due to bone marrow morphology and immunophenotyping (met the WHO 2016 diagnosis criterion) with history of myeloid neoplasms ;
2. Ineligible for allogeneic hematopoietic stem cell transplantation (HSCT) based on local medical standards and clinical decision guidelines in the study;
3. Indications for azacytidine (AZA) treatment were determined according to local medical standards and diagnostic decision guidelines in the study;
4. Morphology and immunophenotyping excluded BCR/ABL positive chronic myelogenous leukemia and other myeloid neoplasms including essential thrombocythemia, polycythemia vera and primary myelofibrosis;
5. Aged 18-80 years old;
6. Alanine transaminase(ALT), Aspartate Transaminase(AST) and serum bilirubin <=2 upper limit of normal (ULN), serum creatinine <=150umol/L, myocardial enzyme <2xULN (of the same age);
7. Left ventricularinjection fraction(LVEF)>=50% by echocardiogram;
8. Estimated glomerular filtration rate (eGFR) ≥30mL/min/1.73m2 ;
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2; 10. must sign (or their legally-acceptable representative must sign) an informed consent form indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. BCR/ABL positive chronic myelogenous leukemia, primary myelofibrosis, polycythemia vera and essential thrombocythemia;
2. Low risk myelodysplastic syndromes according to IPSS or revised IPSS prognostic risk categories;
3. Acute promyelocytic leukemia, myeloid sarcoma, or accelerated or blastic phase of chronic myelogenous leukemia;
4. Allergic to any of the mentioned agent in the study protocol;
5. Pregnant or lactating women, or patients during reproductive stage but not willing to take contraception methods;
6. With obvious dysfunction of liver or kidney, not fulfilling the inclusion criteria;
7. With organic heart disease, which causes clinical symptoms or cardiac dysfunction ( ≥ Class 2 cardiac disease as defined by the New York Heart Association Functional Classification, NYHA );
8. At the same time suffering from other malignant tumors, with the exception of the following: (1) malignancy treated with curative intent and with no evidence of active disease present for more than 5 years prior to screening; (2) adequately treated lentigo maligna melanoma without current evidence of disease or adequately-controlled non-melanomatous skin cancer (even if less than 3 years prior to screening); (3) adequately treated cervical carcinoma in situ without current evidence of disease (even if less than 3 years prior to screening);
9. Known history of human immunodeficiency virus (HIV) or syphilis, or active infection with Hepatitis B (HBV-DNA positive) or Hepatitis C;
10. Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, or history of myocardial infarction within 6 months prior to first dose with study drug, or any Class 3 or 4 cardiac disease as defined by NYHA;
11. Any concurrent medical condition or disease (eg, active systemic infection) that may interfere with the research procedure or outcome, or that the subject may have a risk to participate in the study;
12. Cannot understand or follow the study protocol;
13. Patients under 12 years old or over 80 years old;
14. Received major surgery within 4 weeks prior to randomization;
15. Participated in other clinical researches at the same time one month before enrollment;
16. Cannot matching suitable cord blood stem cell;
17. Addicted to illegal drugs;
18. Have mental disorders or cognitive disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival rate | From the time of randomization to time for up to 2 years.
  It is measured from the date of randomization to the date of death from any cause; patients not known to have died at least follow-up are censored on the date they were last known to be alive.
complete response rate | from randomization to end of cycle 1-2.
  Complete remission was achieved according to the remission criteria of different diseases Complete remission was achieved according to the remission criteria of different diseases Complete remission was achieved according to the remission criteria of different diseases Complete remission was achieved according to the remission criteria of different diseases complete response rate is achieved according to the remission criteria of different diseases
Hematopoietic function recovery time | From the time of randomization to time for up to 2 years.
  The recovery time of hematopoietic function was defined as the time from the decline of three lineages to the stable hematological response of three lineages

SECONDARY OUTCOMES:
The 2-year overall survival rate | From the time of randomization to time for up to 2 years.
  The 2-year survival rate was calculated as the number of surviving cases/the total number of cases followed up for 2 years
disease-free survival | From the time of randomization to time for up to 2 years.
  The disease-free survival was calculated as the time from randomization to disease recurrence or death due to disease progression
Early mortality | up to 3 months
  Early mortality was defined as death within the first 3 months after initiation of induction therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No